CLINICAL TRIAL: NCT03109132
Title: Comfort Check of CO2 Monitoring Cannulas With Oxygen Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: Institute for Skin Research, Israel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: MDT17070
Record Dates: First submitted 2017-01-26; First posted 2017-04-12 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Wearing Comfort

STUDY DESIGN:
Intervention Model Description: This is randomnized crossover study. Every subject will assess all cannulas in randomized order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, order randomized study. All cannulas will be numbered. The investigators, the outcomes assessors and the subjects will be blind to the identity of the cannulas. The order of which the subjects will assess the cannulas will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Model 1 (Active Comparator): Device - O2/CO2 Oral/Nasal cannula sample line - Oridion smart CapnoLine® H Plus with Wedge cannula
  Interventions: Device: Oridion Smart CapnoLine® H Plus with Wedge cannula
- Model 2 (Active Comparator): Device -O2/CO2 Oral/Nasal cannula sample line- Oridion smart CapnoLine® Plus with Non-Wedge cannula
  Interventions: Device: Oridion Smart CapnoLine® Plus with Non-Wedge cannula
- Model 3 (Active Comparator): Device - Experimental sample line Model 3
  Interventions: Device: Experimental sample line Model 3
- Model 4 (Active Comparator): Device - Experimental sample line Model 4
  Interventions: Device: Experimental sample line Model 4
- Model 5 (Active Comparator): Device - Experimental sample line Model 5
  Interventions: Device: Experimental sample line Model 5
- Model 6 (Active Comparator): Device - O2/CO2 cannula w/female luer (Westmed comfort plus #0504)
  Interventions: Device: O2/CO2 cannula w/female luer (Westmed comfort plus #0504)

INTERVENTIONS:
Device: Oridion Smart CapnoLine® H Plus with Wedge cannula — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 1
  Arms: Model 1
Device: Oridion Smart CapnoLine® Plus with Non-Wedge cannula — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 2
  Arms: Model 2
Device: Experimental sample line Model 3 — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 3
  Arms: Model 3
Device: Experimental sample line Model 4 — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 4
  Arms: Model 4
Device: Experimental sample line Model 5 — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 5
  Arms: Model 5
Device: O2/CO2 cannula w/female luer (Westmed comfort plus #0504) — The subjects will assess the comfort level of the different cannulas
  Other Names: Usability test for arm 6
  Arms: Model 6

SUMMARY:
The purpose of this test is to evaluate the comfort level of several model configurations of the Smart CapnoLine plus cannula The test focuses on the comfort / discomfort generated by the device, mainly due to tubes around the ears and on the face skin, the cannula itself (especially in the nostrils and the mouth surrounding) and the smell.

DETAILED DESCRIPTION:
This test compares 4 models for the duration of up to 3 days each and 2 models with duration of up to 24 hours. Each subject will tested the models and will provide feedback at predefined times during the test. During the test and according to initial result the team may decide to shorten the test duration.

The testing staff will include a dermatologist and a technical representative that will supervise the test in order to monitor and control the required performance of the subjects according to test protocol, and relevant outcomes. During the test the dermatologist will monitor any unexpected skin reaction or patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Men and Women
* Age 50-85
* Willingness to participate in the study

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects with sensitivity to any of the products or the its ingredient
* Subjects with sensitivity to preparation for testing bacterial plaque
* Subjects who are treated with anti inflammatory antihistamine corticosteroids treatment
* Subjects who are treated with Anti-thrombotic agents

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Comfort evaluation using self introduction questionnaire | 3 months
  Measuring comfort on a scale of 1 -7, where 1 = not comfortable, 7 = very comfortable Data will be reported using self introduction questionnaires in different time intervals

SECONDARY OUTCOMES:
Comfort evaluation using self introduction questionnaire - calculations | 3 months
  The average comfort will be calculated for each time interval and for the all period. The values has no units, this is a subjective evaluation and not clinical value measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Brenner, Prof., Principal Investigator — The Israeli Institute for Skin Research
Locations (1):
- The Israeli Institute for skin reaserch, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No